CLINICAL TRIAL: NCT06366529
Title: Explore the Value of New Magnetic Resonance Technology in Non-invasive Quantitative Assessment of Renal Dysfunction and Renal Fibrosis
Brief Title: Explore New Magnetic Resonance Technology in Assessment of Renal Dysfunction
Status: Recruiting | Type: Observational
Sponsor: Zhen Li (Other)
Responsible Party: Sponsor-Investigator, Zhen Li, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202308123
Record Dates: First submitted 2024-04-08; First posted 2024-04-16 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Currently, renal biopsy is the gold standard for evaluating renal pathology and renal fibrosis, but it is invasive and carries the risk of serious complications; and the sampled tissue is only a small part of the kidney, which is prone to sampling bias. The lack of reliable, comprehensive test results has hindered the research of new anti-fibrotic drugs and delayed the clinical application of effective new drugs. Therefore, the development of a non-invasive dynamic detection method for renal insufficiency and renal fibrosis in vivo is an urgent clinical problem to be solved.

With the continuous development and update of technology, imaging provides a new way to non-invasively evaluate renal fibrosis. Due to the high resolution of soft tissue and the ability to perform multi-parameter analysis, magnetic resonance has developed the diagnosis of renal insufficiency and renal fibrosis from macroscopic simple biomorphological changes to microscopically complex pathophysiological changes. Many imaging techniques measure renal dysfunction and renal fibrosis by assessing the impact of fibrosis on the functional status, physical properties, and molecular properties of the kidney.

In recent years, in the context of precision medicine, artificial intelligence technologies such as radiomics and machine learning are rapidly becoming very promising auxiliary tools in the imaging assessment of renal fibrosis. It can extract and learn features in images with high throughput, make greater use of information in medical images that cannot be recognized by the human eye, and achieve disease diagnosis, prognosis assessment, and efficacy prediction by building models. However, most of the current research is in the preliminary stage, and there are still few studies on the assessment of renal insufficiency and renal fibrosis. I believe that with the continuous improvement of algorithms and the optimization of models, the progress of radiomics and machine learning will be great. To a certain extent, it promotes the development of personalized medicine and precision medicine for patients with renal insufficiency and renal fibrosis.

DETAILED DESCRIPTION:
Renal insufficiency can be divided into acute kidney injury (AKI) and chronic kidney disease (CKD). There are many causes of AKI, which are mainly divided into three categories: prerenal, renal and postrenal according to the anatomical location. The incidence rate of AKI is about 3% to 10%, and the incidence rate in intensive care units is higher, as high as 30% to 60%; when AKI patients are seriously ill, the mortality rate is higher, about 30% to 80%. The prognosis of AKI is mainly related to the cause and severity of complications. For AKI caused by pre-renal and post-renal causes, if diagnosed early and treated promptly, most patients can recover well in renal function. For patients with AKI caused by renal parenchymal disease, the degree of recovery varies depending on the cause, and some patients will have chronic renal damage. When the duration of AKI is greater than or equal to three months, it can be called CKD. More than 700 million people worldwide suffer from kidney disease, and CKD is the third leading cause of death after tumors and heart disease . CKD can be caused by a variety of kidney diseases, such as diabetic nephropathy, hypertensive nephropathy, and chronic glomerulonephritis. In addition, there is a special type of renal transplant insufficiency, which refers to the renal insufficiency that occurs after a patient undergoes a kidney transplant.

In recent years, people have gradually paid more and more attention to the relationship between various metabolic diseases and body composition analysis and renal insufficiency. These are all risk factors for renal insufficiency. Early identification and management of these risk factors is of great significance to the prognosis and delaying disease progression in patients with renal insufficiency. Over the past 40 years, global obesity rates have continued to rise, with more than one-third of countries having their rates doubled. Moreover, obesity is related to various mechanisms such as insulin resistance, and obese patients are also more likely to suffer from various metabolic diseases. Therefore, obesity is also a factor in renal insufficiency that needs to be prevented and managed urgently. There are anatomical, cellular, and molecular differences in adipose tissue in different parts of the human body. Therefore, it is of great significance to more accurately measure and divide adipose tissue and muscle in the human body and explore its correlation with renal insufficiency. Various metabolic diseases have a high incidence rate, long course, affect tissues and organs throughout the body, and are important risk factors and causes of renal insufficiency. Therefore, it is also important to explore their correlation with renal insufficiency and explore related mechanisms. Contribute to doctors' clinical diagnosis and subsequent auxiliary designation of treatment plans.

However, regardless of its pathogenesis, renal fibrosis is the final pathological manifestation of CKD. Its main pathological characteristics are inflammatory cell infiltration, fibroblast proliferation, extracellular matrix (ECM) deposition, and replacement of normal kidney tissue by scar tissue. Renal fibrosis is the main determinant of renal insufficiency, and its presence and extent are closely related to CKD disease progression and prognosis. Early diagnosis and accurate assessment of the degree of renal insufficiency and renal fibrosis are effective means of delaying the development of end-stage renal disease and are of great clinical significance in improving the survival rate and quality of life of patients with renal insufficiency.

Usually, the indicator used clinically to evaluate renal function is the estimated glomerular filtration rate (eGFR), as well as urea, creatinine, uric acid and bicarbonate to assist in the evaluation. However, these indicators are easily affected by many factors such as drugs and diet, are not very accurate, and may change significantly in a short period of time. More importantly, these indicators reflect overall kidney function. When patients have mild kidney damage and are in the early stages of kidney disease, these indicators are usually still within the normal range. By the time they are significantly reduced, patients have usually developed irreversible kidney damage. The Gates method of renal dynamic imaging is currently the only method widely used in clinical practice to evaluate renal function. However, its examination time is long (more than half an hour), the price is high, and it also imposes a radiation dose on the patient, which limits its routine clinical application.Currently, renal biopsy is the gold standard for evaluating renal pathology and renal fibrosis, but it is invasive and carries the risk of serious complications; and the sampled tissue is only a small part of the kidney, which is prone to sampling bias. The lack of reliable, comprehensive test results has hindered the research of new anti-fibrotic drugs and delayed the clinical application of effective new drugs. Therefore, the development of a non-invasive dynamic detection method for renal insufficiency and renal fibrosis in vivo is an urgent clinical problem to be solved.

With the continuous development and update of technology, imaging provides a new way to non-invasively evaluate renal fibrosis. Due to the high resolution of soft tissue and the ability to perform multi-parameter analysis, magnetic resonance has developed the diagnosis of renal insufficiency and renal fibrosis from macroscopic simple biomorphological changes to microscopically complex pathophysiological changes. Many imaging techniques measure renal dysfunction and renal fibrosis by assessing the impact of fibrosis on the functional status, physical properties, and molecular properties of the kidney. For example, diffusion weighted imaging (DWI) can detect the renal fibrosis process. Changes in the movement of water molecules caused by deposition of extracellular matrix components, infiltration of inflammatory cells and fibroblasts, and renal tubular atrophy; arterial spin labeling (ASL) imaging can detect changes in microvascular perfusion; blood oxygen level dependence (blood oxygen level) oxygenation level-dependent (BOLD) imaging can detect the decrease in tissue oxygenation levels caused by vascular occlusion; magnetic resonance elastography (MRE) can detect the increase in kidney tissue stiffness caused by fibrosis; magnetization transfer imaging, MT) can detect the content of macromolecules such as collagen, etc.

In recent years, in the context of precision medicine, artificial intelligence technologies such as radiomics and machine learning are rapidly becoming very promising auxiliary tools in the imaging assessment of renal fibrosis. It can extract and learn features in images with high throughput, make greater use of information in medical images that cannot be recognized by the human eye, and achieve disease diagnosis, prognosis assessment, and efficacy prediction by building models. However, most of the current research is in the preliminary stage, and there are still few studies on the assessment of renal insufficiency and renal fibrosis. I believe that with the continuous improvement of algorithms and the optimization of models, the progress of radiomics and machine learning will be great. To a certain extent, it promotes the development of personalized medicine and precision medicine for patients with renal insufficiency and renal fibrosis.

This study aims to explore the value of new imaging technologies in the evaluation of patients with renal insufficiency and renal fibrosis, including transplanted renal insufficiency. By obtaining clinical, imaging, laboratory examination and pathological data of patients with renal insufficiency and renal fibrosis, we will use Image processing software analyzes images to explore the relationship between image parameters, body composition and metabolic diseases and the degree of renal insufficiency and renal fibrosis in patients to achieve non-invasive diagnosis, efficacy evaluation and prognosis prediction of renal insufficiency and renal fibrosis. etc., thereby guiding clinical treatment and improving the survival rate and quality of life of patients with renal insufficiency.

Research steps

1. Collection of imaging data: Include patients with the above criteria, communicate with them and make them informed before signing an informed consent form. It is recommended that for MR examinations prescribed by the attending physician, patients should fast for 8 hours and water for 4 hours before the examination. After the examination, the patient's imaging data information should be organized, and information such as image ID and examination item type should be recorded.
2. Image data processing: Use the PACS system and GE workstation to copy the image data in DICOM format, use image processing software to conduct qualitative and quantitative analysis, and record relevant parameter values.
3. Clinical data collection: Query the list of patients through the Radiation Information System (RIS) of the Radiology Department of Tongji Hospital, and collect clinical data, laboratory test data such as serum creatinine, glomerular filtration rate eGFR, etc., and pathological data such as the degree of renal fibrosis. conduct case screening based on the exclusion criteria of this study, and record the patient's medical history in detail, including gender, age, height, weight, blood pressure, past medical history, etc., and laboratory test data including blood routine, blood biochemistry, creatinine, urea, and uric acid. , bicarbonate, glomerular filtration rate eGFR, urinary protein, urinary protein to creatinine ratio, etc., pathological data, pathological type, classification and grading score, renal fibrosis degree score, etc. The treatment situation includes treatment plan, medication, treatment time, etc., Disease follow-up information and other information.
4. Group patients with renal insufficiency and renal fibrosis through laboratory test data such as serum creatinine, glomerular filtration rate eGFR, etc., pathological data such as renal fibrosis degree or score, or treatment efficacy, and compare the groups. Differences in relevant imaging parameters, exploring the ability of different imaging technologies to evaluate renal insufficiency and renal fibrosis, aiming to realize the application of imaging in non-invasive diagnosis, efficacy evaluation, and prognosis prediction of renal insufficiency and renal fibrosis, thereby guiding clinical practice decision making.

7. Possible risks and preventive measures

Possible risks:

This study requires access to patient imaging examination data and electronic medical record data, and there may be risks of leakage of patient privacy and other information.

Precautions:

The imaging data and electronic medical record data used in this study are all data stored by the hospital, which can only be viewed by medical workers except the patients themselves and are used to guide the diagnosis and treatment of diseases and are not used for any commercial activities. The data recorded and used by this institute (including imaging images) do not contain any identifier that can identify the patient. Therefore, the patient's personal information can be effectively protected.

8. Data collection and statistical analysis The data are mainly image parameters analyzed by image processing software. After completing the collection of clinical information, laboratory data, and prognostic data, they are sorted according to the grouping situation and analyzed using statistical software such as SPSS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinically suspected or confirmed renal insufficiency and prescribed MR examination;
2. Age/gender: no limit;
3. Patients who voluntarily participate in clinical trials and sign written informed consent forms

Exclusion Criteria:

1. Patients with pacemakers of unknown material, metal implants in the body, neurostimulators, and claustrophobia, etc.
2. Patients who cannot tolerate sufficient breath-holding for adequate MR examination

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute kidney injury (AKI) and chronic kidney disease (CKD), including patients with renal transplant insufficiency
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
ESKD | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  The patient reaches CKD stage 5 and the glomerular filtration rate is less than 15 ml/min

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital, NO.1095 jiefang avenue, Wuhan, Hubei, China